CLINICAL TRIAL: NCT00939016
Title: The Influence of Dietary Restraint, Social Desirability and Food Type on Accuracy of Reported Dietary Intake
Brief Title: The Influence of Factors on Accuracy of Reported Dietary Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: University of TN IRB 7701 B
Record Dates: First submitted 2009-07-08; First posted 2009-07-14 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Dietary Assessment; 24-hour Dietary Recall; Dietary Restraint; Social Desirability
Keywords: Dietary Assessment; 24-hour dietary recall; Dietary Restraint; Social Desirability; Portion estimation; Underreporting
MeSH Terms: conditions — Social Desirability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- High SD/ Low DR (Active Comparator): This group contains females that exhibit characteristics of high social desirability and low dietary restraint.
  Interventions: Other: Lunch meal with 24 hour dietary recall
- High SD/ High Dr (Active Comparator): This group contains females that exhibit characteristics of high social desirability and high dietary restraint.
  Interventions: Other: Lunch meal with 24 hour dietary recall
- Low SD/ High DR (Active Comparator): This group contains females that exhibit characteristics of low social desirability and high dietary restraint.
  Interventions: Other: Lunch meal with 24 hour dietary recall
- Low SD/ Low DR (Active Comparator): This group contains females that exhibit characteristics of low social desirability and low dietary restraint.
  Interventions: Other: Lunch meal with 24 hour dietary recall

INTERVENTIONS:
Other: Lunch meal with 24 hour dietary recall — Each participant will come into the laboratory for a buffet-style lunch meal, where they are instructed to sample each of the foods served. On the next day, a 24 hour dietary recall is performed to test the participants ability to accurately report amounts and types of food consumed. Measures of dietary restraint and social desirability are taken prior to the laboratory meal via phone interview.

SUMMARY:
The purpose of this study is to evaluate the influence of dietary restraint, social desirability, and food type on the accuracy of dietary intake reported during a 24-hour recall.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the influence of the interaction among dietary restraint, social desirability, and food type ("healthy" vs. "unhealthy") on the accuracy of reporting consumption of a laboratory meal during a 24-hour dietary recall. The automated multiple-pass method (AMPM) of 24-hour dietary recall is considered the gold standard of dietary assessment however the potential for error and biases is widely acknowledged with a tendency towards underreporting. Underreporting has been linked to many factors including two individual characteristics, dietary restraint and social desirability. Both dietary restraint and social desirability have been extensively studied however the influence of their interaction on reported dietary intake is not fully understood. In addition, a relationship to the types of foods (healthy vs. unhealthy) has also been found. For this study, 40 normal-weight female participants will be recruited at The University of Tennessee using flyers inviting volunteers. Participants will be categorized by dietary restraint, high or low, and social desirability, high or low, based on questions during the initial screening. In a laboratory setting participants will consume a meal of pre-weighed foods, including both "healthy" and "unhealthy" foods. The following day, an AMPM 24-hr dietary recall will be conducted with the participant over the telephone. Accuracy of the reported dietary intake of the laboratory meal will be determined by the equation [(reported intake - measured intake)]/measured intake] x100 for amount (weight or volume) and energy (kilocalories) with comparisons between groups and within food types using mixed factorial analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight status (BMI 18.5-24.9)
* Willing to sample study foods

Exclusion Criteria:

* Individuals majoring in Nutrition or Exercise Science
* Smokers
* Individuals taking medication for ADHD
* Individuals who are pregnant
* Individuals with allergies to food in study

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of reported dietary intake compared to measure intake of a laboratory meal. | 1 day.

SECONDARY OUTCOMES:
Dietary Restraint Score of participant. | 1 day.
Social Desirability Score of participant. | 1 day.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, Ph.D., Study Chair — University of Tennessee, Knoxville
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States